CLINICAL TRIAL: NCT04374032
Title: An Open-label, Prospective, Randomized, Comparative Clinical Trial to Evaluate the Efficacy and Safety of ENKORTEN® as an Immunomodulatory Therapy, Within the Usual Therapeutically Established Protocol, for the Treatment of Patients With Moderate to Severe COVID-19 Infection
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of an Immunomodulatory Therapy for the Treatment of Patients With Moderate to Severe COVID-19 Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bosnalijek D.D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN-COVCS-01
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — Enkephalin, Methionine

STUDY DESIGN:
Intervention Model Description: Open-label, prospective, randomized, comparative, multiple doses applied in addition to the standard of care treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENKORTEN (Experimental)
  Interventions: Drug: metenkefalin + tridecactide
- The standard of care treatment (Other): The usual therapeutically established protocol for the treatment of patients with moderate to severe COVID-19 infection
  Interventions: Drug: The standard of care

INTERVENTIONS:
Drug: metenkefalin + tridecactide — ENKORTEN® 5 mg + 1 mg Lyophilisate for Solution for Injection
  Arms: ENKORTEN
Drug: The standard of care — The usual therapeutically established protocol, for the treatment of patients with moderate to severe COVID-19 infection prescribed by The Agency for medicinal products and medical devices of Bosnia and Herzegovina
  Arms: The standard of care treatment

SUMMARY:
An Open-label, prospective, randomized, comparative, multiple doses applied in addition to the standard of care treatment of patients with moderate to severe COVID-19 infection

DETAILED DESCRIPTION:
The justification for the use of immunomodulatory therapy is based on the evidence that drugs that are inhibitors of interleukin IL6 may prevent the more severe lung tissue damage caused by cytokine release in patients with more severe COVID19. Several studies have suggested a "cytokine storm" caused by the release of IL-6, IL-1, IL-12 and IL-18 with tumor necrosis factor TNF alpha and other inflammatory mediators. Increased inflammatory response of lung tissue may result in increased gas exchange at the alveolar-capillary level making oxygenation difficult in patients with more severe forms of the disease and the need for mechanical ventilation. In this regard, it is hypothesized that the use of immunomodulatory therapy should have an effect in reducing the lethal outcome, the need for oxygen therapy, and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with laboratory-confirmed (PCR) COVID-19 infection
* Patients with moderate to severe COVID-19 infection
* Hospitalized patients on clinical centers and cantonal hospitals
* Patients with radiology-confirmed pneumonia within the clinical condition of COVID-19 infection including pulmonary opacity
* Patients with a clinical indication for pneumonia: increased body temperature (defined as a value above ≥ 36.6⁰C axillary route, ≥ 37.2°C oral route or ≥ 37.8 °C rectal route), and/or dyspnea, and/or cough, and/or SpO2 <96%
* Patients aged above 18, both genders
* Patients able and willing to understand the study, adhere to all study procedures and sign a written Informed Consent Form (ICF) prior to entering the study or with the assistance of the witness

Exclusion Criteria:

* Patients not COVID-19 positive
* Patients with mild COVID-19 infection
* Patients who are study subjects in another clinical study for another investigational agent for COVID-19
* Patients with malignant hypertension
* Patients with malignant disease and who are treated for malignant diseases in the last 5 years
* Patients with severe liver and kidney insufficiency
* Patients who are receiving therapy with an immunomodulatory or immunosuppressive agent
* Patients aged below 18, female patients who are pregnant or breastfeeding
* Known allergy to study drug or any component thereof
* Use of haloperidol, dopamine antagonists, or nonsteroidal anti-inflammatory drugs, except paracetamol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Time to onset of change in the patient's clinical condition | 21 day
  The time of onset of improvement in the patient's clinical condition will be measured following the clinical objective and subjective signs and radiological indicators.
Safety and tolerability evaluation - treatment-related adverse events will be assessed by CTCAE | 21 day
  At every examination/evaluation, all AEs, whether noticed by investigators and their associates in the trial, or spontaneously reported by the subjects, or given as answer to direct question, must be evaluated by the investigator and reported on case report forms for AE. AE will be recorded in the e-CRF. Three-degree scale will be used for assessment of AE's severity: mild, moderate, severe.

SECONDARY OUTCOMES:
Length of in-hospital stay | 21 day
  To monitor the period of patient's hospitalization
Survival rate | 21 day
  To monitor the survival rate during the hospitalization
Intubation rate | 21 day
  To monitor the intubation frequency during the hospitalization
Proinflammatory markers levels | 21 day
  To monitor the levels of proinflammatory markers during the hospitalization (IL-6)

CONTACTS AND LOCATIONS:
Overall Officials: Rusmir Baljić, PhD, Principal Investigator — Clinical Center University of Sarajevo
Locations (5):
- Bosnia and Herzegovina (5):
  - Clinical Center University of Sarajevo, Sarajevo, Sarajevo Canton
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - University Clinical Hospital Mostar, Mostar
  - Hospital Travnik, Travnik
  - Cantonal Hospital Zenica, Zenica

IPD SHARING:
Plan to Share IPD: Undecided